CLINICAL TRIAL: NCT03389178
Title: Fetal Early Non-invasive Biomarkers of Chronic Maternal Stress During Pregnancy Resulting in Alterations of Infant Cognitive Development
Brief Title: Fetal Biomarkers of Chronic Maternal Stress During Pregnancy
Acronym: FELICITy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, PD Dr. S. M. Lobmaier, Principal Investigator,, Technical University of Munich
Other Study IDs: FELICITy
Record Dates: First submitted 2017-12-22; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Prenatal Stress
Keywords: prenatal stress; fetal autonomic nervous system; multidimensional FHR variability assessment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- stress group (SG): We will identify prospective subjects according with the inclusion criteria of the study, consistent on singleton pregnant women between 18 to 45 years of age in their third trimester (at least 28 weeks gestation). Upon acceptance participants will enter to Phase I-IV.
  Women and participants will be categorized as stressed or controls after scoring the Cohen Perceived Stress Scale-10 (PSS-10). The PSS-10 has been validated in German speaking populations and will be a quick tool for screening stress among prospective subjects. For the purposes of the current study, a participant with a PSS-10 score ≥19 will be categorized as stressed and entered into Phase II. Recruitment will continue until reaching the aimed cohort of n=75 subjects/group.
  Interventions: Diagnostic Test: Cohen Perceived Stress Scale-10 (PSS-10)
- control group (CG): For every consented subject categorized as stressed, the next screened participant matching for maternal and gestational age with a PSS-10 score < 19 will be entered into Phase II as control.
  Recruitment will continue until reaching the aimed cohort of n=75 subjects/group.
  Interventions: Diagnostic Test: Cohen Perceived Stress Scale-10 (PSS-10)

INTERVENTIONS:
Diagnostic Test: Cohen Perceived Stress Scale-10 (PSS-10) — Participants with a PSS-10 score ≥19 will be categorized as stressed and entered into Phase II. For every consented subject categorized as stressed, the next screened participant matching for maternal and gestational age with a PSS-10 score < 19 will be entered into Phase II as control

SUMMARY:
The investigators´ main hypothesis is that prenatal stress (PS)- induced programming during fetal and postnatal development is reflected in epigenetic and autonomic nervous system (ANS) biomarkers which can be harnessed for early detection and follow-up of affected children. By integrating multiple non-invasively obtainable sources of information using novel epigenetic, electrophysiologic and statistical approaches, the trial could yield progress in maternal-fetal medicine, offering a more precise and truly personalized prediction and new possibilities for designing interventions to improve neurodevelopmental outcomes of pregnancy affected by PS.

DETAILED DESCRIPTION:
Rationale:

A cohort of the population of women attending the center of perinatology at the Department of Obstetrics and Gynecology at the Klinikum rechts der Isar of the Technische Universität München (TUM) for having birth will fall in the group of persons with higher perceived stress levels that might concomitantly carry fetuses that show altered sympathetic and vagal activity.

Experimental design:

This study will be conducted at the Department of Obstetrics and Gynecology at the Klinikum rechts der Isar of the Technische Universität München (TUM) a tertiary center of Perinatology of high complexity located in Munich, Germany and that serves about 2000 mothers/newborns per year. TUM obstetricians will identify prospective subjects according with the inclusion criteria of the study, consistent on singleton pregnant women between 18 to 45 years of age in their third trimester (at least 28 weeks gestation) and without a) serious placental alterations; b) fetal malformations; c) maternal severe illness during pregnancy (i.e. preclampsia), d) maternal drug or alcohol abuse, e) preterm birth (less than 37 weeks) and f) Cord blood pH<7,10.

Prospective participants will be referred to attend an informational session, when procedures will be explained, formal enrollment will be completed and the consent forms from the participants themselves and parental consent for their infants will be obtained. These protocols are in strict accordance with the Committee of Ethical Principles for Medical Research from TUM and has the approval of the Ethics Committee of the Hospital " Klinikum rechts der Isar". Upon acceptance participants will enter to Phase I-IV.

Phase I: Screening:

In this initial stage, the investigators will collect demographic information from consented women and participants will be categorized as stressed or controls after scoring the Cohen Perceived Stress Scale-10 (PSS-10). This questionnaire measures the degree to which situations in one's life are appraised as stressful and is a widely used psychological instrument to measure nonspecific perceived stress. The PSS predicts objective biological markers of stress and increased risk for disease among persons with higher perceived stress levels. In particular, PSS scores were used to relate prenatal stress, anxiety, and depressive symptoms as predictors of intention to breastfeed and to examine correlates of perceived stress in pregnant women. Increased maternal prenatal stress, measured as PSS and anxiety, was associated with temperamental variation of young infants and may represent a risk factor for psychopathology later in life. The PSS-10 has been validated in German speaking populations and will be a quick tool for screening stress among prospective subjects. For the purposes of the current study, a participant with a PSS-10 score ≥19 will be categorized as stressed and entered into Phase II. For every consented subject categorized as stressed, the next screened participant matching for maternal and gestational age with a PSS-10 score < 19 will be entered into Phase II as control. Recruitment will continue until reaching the aimed cohort of n=75 subjects/group.

Phase II: Maternal psychological evaluation and fetal prenatal recordings:

1. Questionnaires: In the context enrolled participants entering this phase will be asked to complete a widely used and validated self-rating questionnaire in order to assess concerns related to pregnancy. The participants will have to complete the Prenatal Distress Questionnaire (PDQ-12) designed to assess specific worries and concerns pertaining to pregnancy and includes items on concerns regarding medical problems, physical symptoms, parenting, relationships, bodily changes, labour and delivery, and the health of the baby. This instrument has been previously applied in numerous studies involving pregnant women from diverse cultural and socio-economic backgrounds and is an effective instrument to assess pregnancy related stress. PDQ-12 has been translated into German and was validated. Additionally participants will fill in a questionnaire about their education level, socio-economic situation, ethnicity and clinical history.
2. ANS assessment: During the same visit the fetal heart rate (FHR) will be measured by a routine cardiotocography (CTG) and simultaneously by transabdominal electrocardiography (transabdominal-fetal ECG). The electrophysiological signal contains the maternal ECG (mECG), fetal ECG (fECG) and noise, it will be recorded using 5 disposable electrodes. The five disposable electrodes will be placed on the maternal abdomen in a standardized manner. Before placing the electrodes, skin impedance will be reduced by using abrading paper at the electrode placement site. Data will be analyzed off line after computer download. For the case that signal loss is high with fECG method, which is a known problem (more frequent between 28 to 32 gestational weeks, but also might occur after that period), conventional external CTG will be performed simultaneous using an ultrasound transducer placed on the maternal Abdomen. The investigators will analyze the impact of PS on ANS activity by deploying advanced methods of FHR monitoring: phase-rectified signal averaging (PRSA), multidimensional FHR variability analysis and assessment of maternal-fetal heart rate synchronization FECG registrations as well as CTG registrations will be performed once during pregnancy for at least 40 minutes to get fetal activity status. During labour conventional CTG and if possible fECG and mECG will be performed simultaneously.

Phase III: Delivery:

1. Maternal cortisol assessment: Cortisol, the hormonal product of activation of the hypothalamic-pituitary-adrenal (HPA) axis has been suggested as a potential mechanism linking maternal stress and perinatal outcome. Single blood and /or saliva samples provides a measure at a single point in time and considering its major physiological daily fluctuations, may not be the most informative measure to evaluate overall or long term HPA activity during the prenatal period. Recently, the use of hair cortisol measurements demonstrated that it provides a retrospective index of integrated cortisol secretion over periods of several months . It is postulated that cortisol is incorporated into the emerging hair and slowly grow with it. Therefore the amount of cortisol in a particular hair segment is assumed to reflect the integrated systemic steroid hormone concentration over a growth period of a specific hair segment. Hair and salivary cortisol are highly correlated in non-human primates and it has been demonstrated increased hair cortisol concentrations in pregnant women. Therefore, hair cortisol has the potential to serve as an integrated measure of HPA activity over an extended period of time of up to 3-6 months. On the day of parturition, hair strands (~3 mm diameter) will be collected from the posterior vertex region on the head as close to the scalp as possible as recommended by the Society of Hair Testing (Soc of Hair testing, 1997). Based on an approximate hair growth rate of 1 cm per month, the proximal 3 cm long hair segment is assumed to reflect the integrated hormone secretion over the three-month-period prior to sampling. The 3 cm hair sample will be wrapped in aluminum foil for protection and stored at room temperature. Hair samples will be sent for cortisol determination.
2. Maternal blood collection (not part of this study- blood will be stored at the biobank): A maximum of 20 ml will be collected to provide serum and plasma specimens. The blood specimens will be stored in 2-4 x 1.8 ml labelled Cryotube vials after one centrifugation cycle for serum specimens (2750 rpm x 10 min at RT) and stored at -80 °C and after 10 gentle invertions for plasma specimens and stored at -20 °C. The blood samples will be processed and frozen within 2-4 h. The time interval between collection and freezing will be recorded for all specimens.
3. Cord Blood samples: Once the baby is delivered and before placental separation, the cord is clamped and cord blood samples will be drawn and distributed in two tubes for serum and plasma specimens following the same procedure as detailed above. A third sample will be collected in a PAXgene tube, carefully inverted 10 times and left at RT for 5 hs in an upright position. The tubes will then be stored at -80 °C after 10-16 hs at -20 °C. (the PAXgene sample is not part of this study- blood will be stored at the biobank)
4. Placenta samples (not part of this study- samples will be stored at the biobank): Once the placenta is delivered the maternal side will be dissected. Two biopsies will be taken (approximately 1 cm³) avoiding decidua contamination. The samples are placed in Cryotube vials and stored immediately at -20 °C.
5. Newborn recordings: Soon after birth, a neonatal specialized midwife will collect a saliva/buccal samples from the newborns by gentle rubbing the gums on both sides with the sponge of the Oracollect-DNA kit (DNA Genotek, Canada) and stored at RT. Clinical data including body metrics pH and APGAR score, will be recorded.

Phase IV: Postnatal recordings:

Following up on the cohort recruited at phase I and mirroring the neurodevelopmental animal study, we will perform a longitudinal study to explore the feasibility of measuring biomarkers of PS-induced epigenetic reprogramming.

1. Infant developmental assessment: In the final stage of the study, the mother will be asked to complete a final questionnaire to assess postpartum depression and breast feeding that she will receive by mail post. While the current study is focused on antenatal events, early postnatal care is heavily impacted by maternal depression and can alter the epigenetic reprogramming of the infant brain. Therefore, the level of maternal involvement in childcare during the first months could directly affect the methylation status and will be recorded. Mothers will be asked about feeding and care routines to complete the postnatal-care assessment.
2. Infants' cognitive development will be assessed by Bayley Scale III of Infant development (BSID) at 18 months of age. The BSID is composed by a series of tests aimed at evaluating cognitive, motor and behavioral development on infants from age 0-3 years. The Mental Development Index and the Psychomotor Development Index components have a mean score of 100 and a standard deviation of 15 (range of 55 to 145). Scores between 70-84 indicate mildly delayed performance, and scores ≤ 69 indicate significantly delayed performance. Approximately 13.5 % of tested infants are expected to fall in those categories. Maternal psychological distress during pregnancy was associated in a dose-response manner with BSID scores in 2 years-old children. A specialized Psychologist, who will be blind regarding maternal stress categorization, will administer the tests, which will last about 40 minutes.
3. A new saliva sample will be collected from the infants at this final visit. The biomarkers will be quantified from salivary DNA obtained from the young infants. ECG will be measured for ANS assessment. Methylation levels will be correlated with maternal stress, depression and anxiety, with infant's cognitive development and ANS capacity to assess the efficacy of these novel biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnant women between 18 to 45 years of age in their third trimester (at least 28 weeks gestation)

Exclusion Criteria:

* serious placental alterations;
* fetal malformations;
* maternal severe illness during pregnancy (i.e. preclampsia),
* maternal drug or alcohol abuse,
* preterm birth (less than 37 weeks) and
* Cord blood pH<7,10.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: A cohort of the population of women attending the center of perinatology at the Department of Obstetrics and Gynecology at the Klinikum rechts der Isar of the Technische Universität München (TUM) for having birth will fall in the group of persons with higher perceived stress levels that might concomitantly carry fetuses that show altered sympathetic and vagal activity.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
fetal hear rate (FHR) signatures | 12 months
  The impact of prenatal stress (PS) on autonomic nervous system (ANS) activity will be analyzed by deploying advanced methods of FHR monitoring: phase-rectified signal averaging (PRSA), multidimensional FHR variability analysis and assessment of maternal-fetal heart rate synchronization. We expect that children affected by PS show early alterations of fetal ANS.
methylation levels by Epigenome-Wide Association Study (EWAS) | 12 months

SECONDARY OUTCOMES:
neuro development at 18 months of age | 18 months after birth
  Infants' cognitive development will be assessed by Bayley Scale III of Infant development (BSID) at 18 months of age. The BSID is composed by a series of tests aimed at evaluating cognitive, motor and behavioral development on infants from age 0-3 years. The Mental Development Index and the Psychomotor Development Index components have a mean score of 100 and a standard deviation of 15 (range of 55 to 145). Scores between 70-84 indicate mildly delayed performance, and scores ≤ 69 indicate significantly delayed performance. Approximately 13.5 % of tested infants are expected to fall in those categories. Maternal psychological distress during pregnancy was associated in a dose-response manner with BSID scores in 2 years-old children. A specialized Psychologist, who will be blind regarding maternal stress categorization, will administer the tests.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Lobmaier, MD, PhD, Principal Investigator — Frauenklinik, Klinikum rechts der Isar, Technical University of Munich
Locations (1):
- Klinikum rechts der Isar, München, Bavaria, Germany

REFERENCES:
- [Derived] Sharma R, Frasch MG, Zelgert C, Zimmermann P, Fabre B, Wilson R, Waldenberger M, MacDonald JW, Bammler TK, Lobmaier SM, Antonelli MC. Maternal-fetal stress and DNA methylation signatures in neonatal saliva: an epigenome-wide association study. Clin Epigenetics. 2022 Jul 14;14(1):87. doi: 10.1186/s13148-022-01310-x. PMID 35836289
- [Derived] Lobmaier SM, Muller A, Zelgert C, Shen C, Su PC, Schmidt G, Haller B, Berg G, Fabre B, Weyrich J, Wu HT, Frasch MG, Antonelli MC. Fetal heart rate variability responsiveness to maternal stress, non-invasively detected from maternal transabdominal ECG. Arch Gynecol Obstet. 2020 Feb;301(2):405-414. doi: 10.1007/s00404-019-05390-8. Epub 2019 Nov 28. PMID 31781889